CLINICAL TRIAL: NCT03973840
Title: A Study to Assess Post-collection Conversion of Testosterone Undecanoate (TU) to Testosterone in Blood From Men Receiving Oral TU Collected Into Different Types of Sample Tubes
Brief Title: Assessment of Blood From Men Receiving Oral TU in Various Collection Tubes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Clarus Therapeutics, Inc. (Industry)
Collaborators: Celerion; Syneos Health; ARUP Laboratories (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CLAR-18019
Record Dates: First submitted 2019-06-02; First posted 2019-06-04 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Hypogonadism, Male
MeSH Terms: conditions — Eunuchism | interventions — testosterone undecanoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- healthy men treatment arm (Experimental): Subjects were given 15 doses over 8 days, and then blood was drawn into several types of collection tubes at different storage conditions.
  Interventions: Drug: Testosterone Undecanoate

INTERVENTIONS:
Drug: Testosterone Undecanoate — dose was given orally and allowed to reach steady state

SUMMARY:
To describe the rate of post-collection TU to testosterone conversion, as manifested by increases in testosterone concentration, in Plain tubes held at room temperature and sodium fluoride (NaF)-ethylenediaminetetraacetic acid (EDTA) tubes held at room temperature or on ice prior to centrifugation

DETAILED DESCRIPTION:
This was an open-label, non-randomized, single-sequence study in which men dosed with JATENZO had blood drawn into 3 different types of blood-collection tubes (ie, Plain, EDTA, and NaF-EDTA). These tubes were then processed in different ways (ie, different durations between phlebotomy and centrifugation, different holding temperatures [room temperature or on ice] between phlebotomy and centrifugation). After defined periods of incubation, the tubes were centrifuged and the serum/plasma transferred into vials and frozen. The testosterone and TU levels in the serum/plasma were then measured using validated liquid chromatography/tandem mass spectrometry assays.

ELIGIBILITY:
Inclusion Criteria:

Subjects were required to meet all of the following criteria in order to be eligible for the study:

1. Male (gender at birth) 18 to 65 years of age, inclusive, and legally able to give informed consent, as applicable by law. The percentage of non-Hispanic and Hispanic men was specified to be approximately ≥ 70% and ≤ 30%, respectively.
2. Adequate venous access in the left or right arm to allow collection of a number of blood samples via a venous cannula or needle sticks
3. Naïve to androgen-replacement therapy
4. Willing to consume the entire protocol-specified breakfast and dinner meals
5. Average screening systolic blood pressure < 140 mmHg and/or diastolic blood pressure < 90 mmHg
6. Voluntarily gave written informed consent to participate in this study -

Exclusion Criteria:

Subjects who met any of the following criteria were not eligible for participation in this study:

1. History of hypertension or taking anti-hypertensive medications
2. Intercurrent disease deemed clinically significant, in the opinion of the Investigator, of any type; in particular, liver, kidney, uncontrolled or poorly controlled heart disease, including congestive heart failure, coronary heart disease, heart attack or cerebrovascular accident in prior 6 months, or psychiatric-illness, including severe depression
3. Electrocardiogram which Principal Investigator, or designate, believed was clinically significantly abnormal
4. Intercurrent process or disease which could have impacted the absorption of JATENZO, in particular vomiting, nausea, diarrhea, or inflammatory bowel disease
5. Current use of the following groups of drugs that affect testosterone levels, testosterone metabolism, or levels of testosterone metabolites, namely antiandrogens, 5 alpha reductase inhibitors (eg, dutasteride, finasteride), estrogens, long-acting opioid analgesics (eg, methadone hydrochloride, buprenorphine hydrochloride), or human growth hormone
6. History of or was currently being evaluated for breast or prostate cancer
7. Prostate specific antigen above the upper limit of normal
8. Positive test for antibodies to human immunodeficiency virus type 1 or 2, hepatitis B surface antigen, or antibodies to hepatitis C virus at the Screening visit
9. Positive urine drug test at the Screening visit
10. Current treatment with oral lipase inhibitors (eg, orlistat [Xenical]), bile acid-binding resins (eg, cholestyramine [Questran], colestipol [Colestid]), fibric acid derivatives (eg, clofibrate [Atromid-X], gemfibrozil [Lopid]), and probucol (Lorelco).
11. Smokers who were unable to refrain from smoking during the confinement period required in this study
12. Current evidence of or history of abuse of alcohol or any drug substance within the previous 2 years
13. Receipt of any drug as part of a research study within 30 days of initial dose administration in this study
14. Blood donation (usually 550 mL) within the 12-week period before the initial study drug dose
15. Hematocrit < 35% or > 50%
16. Body mass index ≥ 31 kg/m2 -

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
measure rate of post-collection TU-to-testosterone conversion in 3 types of collection tubes | 8 days
  To describe the rate of post-collection TU to testosterone conversion, as manifested by increases in testosterone concentration, in Plain tubes held at room temperature and sodium fluoride (NaF)-ethylenediaminetetraacetic acid (EDTA) tubes held at room temperature or on ice prior to centrifugation

SECONDARY OUTCOMES:
rate of post-collection TU-to-testosterone conversion, as manifested by increases in testosterone concentration, in EDTA and NaF-EDTA collection tubes | 8 days
  To describe the rate of post-collection TU to testosterone conversion, as manifested by increases in testosterone concentration, in EDTA and NaF-EDTA tubes held at room temperature or on ice prior to centrifugation
magnitude of overestimation of the true circulating testosterone concentration at 5 hours postdose | 8 days
  To estimate the magnitude of overestimation of the true circulating testosterone concentration at 5 hours postdose, when blood was collected in various tubes and the tubes were held at room temperature or on ice.
healthy men's testosterone levels in serum and plasma | 8 days
  To compare healthy men's testosterone levels in serum and plasma from Plain and EDTA tubes, respectively

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 8 days
  To characterize the safety and tolerability of JATENZO

CONTACTS AND LOCATIONS:
Locations (1):
- Clarus Therapeutics, Inc, Northbrook, Illinois, United States

IPD SHARING:
Plan to Share IPD: No